CLINICAL TRIAL: NCT00220194
Title: A Six-Month, Open-Label, Crossover Study Of the Maintenance Of Serum Testosterone And PSA Suppression After Switching Between Lupron 22.5 Mg And Eligard 22.5 Mg Or Zoladex 10.8 Mg And Eligard 22.5 Mg In Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: San Bernardino Urological Associates Medical Group Inc (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SBU001; Sanofi Aventis
Record Dates: First submitted 2005-09-17; First posted 2005-09-22 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Cancer of Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide

INTERVENTIONS:
Drug: leuprolide acetate

SUMMARY:
Comparing the effect of switching from Lupron and Zoladex to Eligard. PSA and Testosterone levels are measured at set intervals to determine if Eligard is equal or better then Lupron or Zoladex in advanced Prostate Cancer patients.

ELIGIBILITY:
Inclusion Criteria: Patient with Advanced Ca, on stable dose of Lupron or Zoladex

-

Exclusion Criteria:

* Previous exposure to Eligard.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-04; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Franklin M Chu, MD, Principal Investigator — San Bernfardino Urological Associates
Locations (1):
- San bernardino Urological Associates Medical Group, San Bernardino, California, United States